CLINICAL TRIAL: NCT02106078
Title: 2/2-A Randomized Trial of Internet-Based Interventions for Bipolar Disorder
Brief Title: Internet-Based Interventions for Bipolar Disorder
Acronym: MoodSwings 2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: VA Palo Alto Health Care System (U.S. Federal Agency)
Collaborators: University of Melbourne (Other)
Responsible Party: Principal Investigator, patricia suppes, Director, Bipolar and Depression Research Program, VA Palo Alto Health Care System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1R34MH091284 (NIH)
Record Dates: First submitted 2013-05-16; First posted 2014-04-07 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2015-09

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder; Bipolar; Online Intervention; Internet intervention; Self-Help
MeSH Terms: conditions — Bipolar Disorder | interventions — Self-Help Groups; Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Level 1 (Active Comparator): Moderated discussion board only
  Interventions: Behavioral: Moderated Discussion Board
- Level 2 (Active Comparator): Moderated discussion board plus psychoeducation
  Interventions: Behavioral: Moderated Discussion Board; Behavioral: Psychoeducation
- Level 3 (Active Comparator): Moderated discussion board plus psychoeducation plus interactive psychosocial tools
  Interventions: Behavioral: Moderated Discussion Board; Behavioral: Psychoeducation; Behavioral: Interactive Psychosocial Tools

INTERVENTIONS:
Behavioral: Moderated Discussion Board — All groups will have access to asynchronous, moderated discussion boards. Assignment to discussion board will be stratified by randomization group (Level 1, 2 or 3). Level 1 access to the discussion board will serve as our "peer support" control condition, although we do expect some modest benefit from this intervention alone (Mead et al., 2010).
  The discussion boards will be moderated by trained clinicians (masters level or higher). Discussion boards will be asynchronous, with all posts screened by the moderator(s) before appearing to the group.
  Other Names: discussion board; online discussion; online posts; online discussion boards; forum; discussion forum; support group; discussion group
Behavioral: Psychoeducation — Online psychoeducation is only available to those randomized to Levels 2 and 3. The core modules of MoodSwings 2.0 will use videos and improved organization of content based on feedback from previous pilot work. Module topic areas include:
  1. What is bipolar disorder? - Content about symptoms and diagnosis
  2. Stress and triggers of illness
  3. Medication and the biological basis of bipolar disorder
  4. Depression - Symptoms, early detection and helpful strategies
  5. Mania and hypomania - Symptoms, early detection and helpful strategies
  Other Names: Online psychoeducation; Online education; Education
  Arms: Level 2; Level 3
Behavioral: Interactive Psychosocial Tools — Online psychosocial tools are only available to those randomized to Level 3. They include structured mood monitoring, medication monitoring, and life charting visual tools. There are also interactive worksheets that encourage awareness of negative thoughts and strategies to challenge them, help participants weight the costs and benefits of different behaviors, problem solving and goal setting, and reinforcing self-affirmation. Participants have the opportunity to build a record of personal triggers of illness and illness profile - including early warning signs, and symptoms typically experienced during an episode of illness, as well as a personal "relapse prevention plan."
  Other Names: Interactive tools; Online tools; Online interactive tools
  Arms: Level 3

SUMMARY:
The investigators hope to learn whether access to online support and education can help people with Bipolar Disorder (BD) better manage their symptoms of depression.

DETAILED DESCRIPTION:
This study will examine if there is a benefit of an online intervention for persons with bipolar diagnoses, and what components appear to be useful. Specifically, the study will examine (1) whether exposure to the MoodSwings 2.0 intervention results in decreased depressive symptoms as measured by the Montgomery Asberg Rating Scale for Depression (MADRS) and (2) whether there is an association between graduated levels of involvement (Level I, 2, or 3) and resulting improvement? We expect that those participants assigned to the control condition (Level 1, peer discussion board only), will have fewer positive outcomes than those in Level 2 (discussion board and psychoeducation) or 3 (discussion board, psychoeducation, and interactive psychosocial tools) conditions.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of bipolar I disorder, bipolar II disorder, or bipolar disorder NOS verified with the Structured Clinical Interview for the Diagnostic and Statistical Manual for Mental Disorders (SCID) Mood disorder module.
* Age 21-65.
* Access to a computer with internet access. Access to a printer is preferable, but not required.
* Able to speak and read English proficiently.
* Some degree of medical supervision of bipolar disorder (sees a health professional at least twice a year to discuss symptoms and treatment needs) and local access to emergency care.

Exclusion Criteria:

* Current psychosis, as assessed in screening phone interview with the SCID psychosis module.
* Acutely suicidal (defined as having a HAM-D item 3, score of ≥3).
* Current mania, assessed using mania module of the SCID mood disorders module.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Montgomery Asberg Rating Scale (MADRS) for Depression | Change from Baseline to 3 months, 6 months, 9 months and 12 months
  The MADRS is a 10-item scale, completed by the clinician to assess symptoms of depression. It is particularly sensitive to changes in depression over time. Joint reliability for the total score across several studies ranged from 0.76 to 0.95, and it is viewed as a reliable and valid measure of depression symptoms.
Young Mania Rating Scale | Change from Baseline to 3 months, 6 months, 9 months and 12 months
  The YMRS is an 11-item scale, completed by the clinician to assess symptoms of mania. This scale is viewed as a reliable and valid measure of manic symptoms, and is sensitive to changes in mania over time.

SECONDARY OUTCOMES:
Time to Intervention for Mood Episode( TIME) | Changes from Baseline to 3 months, 6 months, 9 months and 12 months
  Relapse or time to intervention will be assessed using Time Scale , with intervention defined as initiation, discontinuation, or dose adjustment of a treatment, initiation of psychotherapy or ECT, visit to an emergency provider or hospitalization in response to new mood symptoms.
SF-12 | Change from Baseline to 3 months, 6 months, 9 months and 12 months
  The SF-12 is a short, multipurpose measure of perceived impairment due to health problems. It is widely used as a short version of the SF-36, and has good validity. The SF-12 yields two risk-adjusted summary scores, impairment perceived as due to physical illness and impairment perceived as due to emotional problems (Ware et al., 1996)
Cornell Service Index (CSI) | Change from Baseline to 3 months, 6 months, 9 months and 12 months
  Use of general medical and psychiatric health services will be collected via the Cornell Service Index (CSI; Sirey et al., 2005). The CSI is a brief assessment of health service use. It has good inter-rater and test-retest reliability and assesses four types of services: outpatient psychiatric or psychological services (e.g., psychotropic medication visits or psychotherapy), outpatient medical services (e.g., visits to medical providers), professional support services (e.g., home health nurse visits, meal delivery), and intensive services (e.g., emergency department visits or hospitalization).
Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) | Change from baseline to 3 months, 6 months, 9 months and 12 months
  The Quality of Life, Enjoyment and Satisfaction Questionnaire (Q-LES-Q) assesses subjective quality of life(i.e. physical health, subjective feelings, leisure activities and and social relationships). The 16 item short form is designated to measure satisfaction with various areas of daily functioning, such as social relationships, living/housing, physical heath, medication and global satisfaction.
Medication Adherence rating Scale( MARS) | Changes from Baseline to 3 months, 6months, 9 months and 12 months
  When applicable, adherence to prescribed medication will be assessed with the Medication Adherence Rating Scale(MARS). This 10-item scale has acceptable reliability, with Cronbach's alpha.75, and test re-test reliability 0.72. It is seen as a valid measure with significant correlations with other measures of medication adherence(p<.01) and with serum blood levels at p< .05.
Patient satisfaction Questionnaire 18( PSQ-18) | Changes from Baseline to 3 months, 6 months, 9 months and 12 months
  The Patient satisfaction Questionnaire 18 assesses the overall satisfaction of each participant with their current medical care. This 18-item scale is a short form version of the 50-item Patient satisfaction Questionnaire. The PSQ sub-scales show acceptable internal consistency reliability. Furthermore, corresponding PSQ 18 and PSQIII subscales are substantially correlated with one another.
Treatment Satisfaction Questionnaire- Modified | Changes from Baseline to 3 months, 6 months, 9 months and 12 months
  For the purposes of this study, the Treatment satisfaction Questionnaire- Modified was revised to suit the bipolar disorder and the MoodSwings 2.0 Program. This questionnaire was originally a modified version of the Treatment Satisfaction Questionnaire
Medical Outcomes Study Social Support Survey( MOS-SSS) | Changes from Baseline to 3 months, 6 months, 9 months and 12 months
  Social support will be assessed with the Medical Outcomes Study Social Support Survey. This 18-item scale has acceptable reliability( alpha > 0.91) and construct validity, and was specifically developed for people with chronic conditions.

OTHER OUTCOMES:
Inventory Of Stigma Experiences | Changes from Baseline to 3 months, 6 months, 9 months and 12 months
  This scale will be used to measure both the self reported experiences of stigma and the impact of stigma
Motivation for Treatment Questionnaire - 8 item ( MTQ 8) | Changes from Baseline to 3 months, 6 months,9months and 12 months
  The motivation for Treatment Questionnaire( MTQ-8) consists of eight questions to assess motivational reasons to seek treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Suppes, MD, PhD, Principal Investigator — VA Palo Alto Health Care System & Stanford University School of Medicine
Locations (1):
- VA Palo Alto Healthcare System, Palo Alto, California, United States

REFERENCES:
- [Derived] Gliddon E, Cosgrove V, Berk L, Lauder S, Mohebbi M, Grimm D, Dodd S, Coulson C, Raju K, Suppes T, Berk M. A randomized controlled trial of MoodSwings 2.0: An internet-based self-management program for bipolar disorder. Bipolar Disord. 2019 Feb;21(1):28-39. doi: 10.1111/bdi.12669. Epub 2018 Jun 21. PMID 29931798
- [Derived] Gliddon E, Lauder S, Berk L, Cosgrove V, Grimm D, Dodd S, Suppes T, Berk M. Evaluating discussion board engagement in the MoodSwings online self-help program for bipolar disorder: protocol for an observational prospective cohort study. BMC Psychiatry. 2015 Oct 14;15:243. doi: 10.1186/s12888-015-0630-7. PMID 26462799
- See also: MoodSwings Website — http://moodswings.net.au/